CLINICAL TRIAL: NCT00265941
Title: A Randomized Phase III Trial of Concurrent Accelerated Radiation and Cisplatin Versus Concurrent Accelerated Radiation, Cisplatin, and Cetuximab (C225) [Followed by Surgery for Selected Patients] for Stage III and IV Head and Neck Carcinomas
Brief Title: Radiation Therapy and Cisplatin With or Without Cetuximab in Treating Patients With Stage III or Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 0522; CDR0000458049; NCI-2009-00729 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RT + cisplatin (Active Comparator): Radiation therapy (RT) as accelerated fractionation by concomitant boost (AFX-CB) or intensity-modulated radiation therapy (IMRT) plus cisplatin
  Interventions: Drug: cisplatin; Radiation: Accelerated Fractionation by Concomitant Boost; Radiation: Intensity-modulated radiation therapy
- RT + cisplatin + cetuximab (Experimental): Radiation therapy (RT) as accelerated fractionation by concomitant boost (AFX-CB) or intensity-modulated radiation therapy (IMRT) plus cisplatin plus cetuximab
  Interventions: Drug: cetuximab; Drug: cisplatin; Radiation: Accelerated Fractionation by Concomitant Boost; Radiation: Intensity-modulated radiation therapy

INTERVENTIONS:
Drug: cetuximab — Cetuximab 400 mg/m^2 IV loading dose 5-7 days before start of radiation therapy, then 250 mg/m^2 IV weekly for 7 weeks
  Arms: RT + cisplatin + cetuximab
Drug: cisplatin — Cisplatin 100 mg/m^2 IV on days 1 and 22
Radiation: Accelerated Fractionation by Concomitant Boost — 3DCRT 54 Gy in 30 1.8 Gy fractions over 6 weeks with boost 18 Gy in 12 1.5 Gy fractions for last 12 days, for a total of 72 Gy in 42 fractions over 6 weeks
  Other Names: AFX-CB
Radiation: Intensity-modulated radiation therapy — 70 Gy in 35 2.0 Gy fractions over 6 weeks with 6 fractions per week (on Saturday or as second daily fraction) in 5 of the 6 weeks.
  Other Names: IMRT

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Cisplatin may also make tumor cells more sensitive to radiation therapy. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving radiation therapy and cisplatin together with cetuximab may kill more tumor cells. It is not yet known whether radiation therapy and cisplatin are more effective with or without cetuximab in treating head and neck cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy, cisplatin, and cetuximab to see how well they work compared to radiation therapy and cisplatin in treating patients with stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate whether the addition of cetuximab to a concurrent radiation-cisplatin regimen will improve progression-free survival in patients with stage III or IV squamous cell carcinoma of the oropharynx, hypopharynx, or larynx.

Secondary

* Determine the impact of the addition of cetuximab to a concurrent radiation-cisplatin regimen on overall survival, local-regional control, acute and late toxic effects, quality of life, and health utilities in these patients.
* Correlate the expression of epidermal growth factor receptor (EGFR) and its down-stream molecules with outcome in patients participating in this component of the trial.
* Correlate pre-treatment positron emission tomography (PET) scan findings with progression-free survival, overall survival, and local-regional control in patients participating in this component of the trial.
* Correlate post-treatment PET scan findings with nodal response and nodal relapse in patients participating in this component of the trial.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are stratified according to primary site (larynx vs non-larynx), nodal stage (N0 vs N1, N2a, N2b vs N2c, N3), Zubrod performance status (0 vs 1), use of intensity modulated radiotherapy (IMRT) (no vs yes), and pre-treatment PET/CT scan (no vs yes). Patients are randomized to 1 of 2 treatment arms.

NOTE: *A neck dissection is optional for patients with multiple lymph nodes or lymph nodes > 3 cm in diameter who achieve a complete clinical and radiographic response in the neck.

Quality of life is assessed at baseline, once during the last 2 weeks of treatment, at 3 and 12 months from the start of treatment, and then annually for 4 years.

After completion of study treatment, patients are followed periodically for 5 years and then annually thereafter.

ELIGIBILITY:
Inclusion criteria:

* Pathologically (histologically or cytologically) proven (from primary lesion and/or lymph nodes) diagnosis of squamous cell carcinoma of the oropharynx, hypopharynx, or larynx;
* Selected stage III or IV disease (T2N2-3M0, T3-4 any N M0); Note: Patients with T1, any N, or T2N1 tumors are not eligible.
* Appropriate stage for protocol entry, including no distant metastases, based upon the following minimum diagnostic workup:
* History/physical examination within 4 weeks prior to registration, including assessment of weight and weight loss in past 6 months and an examination by a Medical Oncologist;
* Chest x-ray (or Chest CT scan or PET/CT scan) within 6 weeks prior to registration;
* CT scan or MRI of the head and neck (of the primary tumor and neck nodes) or PET/CT scan within 6 weeks prior to registration; see Section 6.11 for details of PET scans. Note: A PET/CT can only be used instead of a CT scan or MRI if the CT is a high quality scan with contrast.
* Left ejection fraction determined by echocardiogram and/or multiple gated acquisition (MUGA) technique within 12 weeks of registration;
* Zubrod Performance Status 0-1;
* Age > 18;
* Adequate bone marrow function, defined as follows:
* Absolute neutrophil count (ANC) > 1,800 cells/mm3 based upon CBC/differential obtained within 2 weeks prior to registration on study;
* Platelets > 100,000 cells/mm3 based upon complete blood count (CBC)/differential obtained within 2 weeks prior to registration on study;
* Hemoglobin > 8.0 g/dl based upon CBC/differential obtained within 2 weeks prior to registration on study (Note: The use of transfusion or other intervention to achieve Hgb > 8.0 g/dl is acceptable.)
* Adequate hepatic function, defined as follows:
* Bilirubin < 1.5 mg/dl within 2 weeks prior to registration on study; For patients with Gilbert's disease as the sole cause of elevated bilirubin, please contact the PI, Dr. Ang.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2x the upper limit of normal within 2 weeks prior to registration on study;
* Adequate renal function, defined as follows:
* Serum creatinine < 1.5 mg/dl within 2 weeks prior to registration
* Creatinine clearance (CCr) ≥ 50 ml/min within 2 weeks prior to registration determined by 24-hour collection or estimated by Cockcroft-Gault formula: CCr male = [(140 - age) x (wt in kg)]/[(Serum Cr mg/dl) x (72)] CCr female = 0.85 x (CrCl male)
* Pregnancy test within 2 weeks prior to registration for women of childbearing potential;
* Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study (until at least 60 days following the last study treatment);
* Patient must sign study specific informed consent prior to study entry.

Exclusion criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years;
* Patients with simultaneous primaries or bilateral tumors are excluded.
* Gross total excision (e.g., by tonsillectomy) of the primary tumor; however, partial removal of the tumor to alleviate an impending airway obstruction does not make the patient ineligible.
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable;
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
* Primary site of tumor of oral cavity, nasopharynx, sinuses, or salivary glands;
* Initial surgical treatment, excluding diagnostic biopsy of the primary site or nodal sampling of neck disease; radical or modified neck dissection is not permitted.
* Severe, active co-morbidity, defined as follows:
* Current uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction;
* Left Ventricular Ejection Fraction < 45%;
* Transmural myocardial infarction within the last 6 months;
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
* Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration;
* Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
* Any uncontrolled condition, which in the opinion of the investigator, would interfere in the safe and timely completion of study procedures;
* CTCAE, v. 3.0 grade 3-4 electrolyte abnormalities:

  * Calcium < 7 mg/dl or > 12.5 mg/dl;
  * Glucose < 40 mg/dl or > 250 mg/dl;
  * Magnesium < 0.9 mg/dl or > 3 mg/dl;
  * Potassium < 3 mmol/L or > 6 mmol/L;
  * Sodium < 130 mmol/L or > 155 mmol/L
* Pregnant or lactating women or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
* Prior allergic reaction to the study drug(s) involved in this protocol;
* Prior therapy that specifically and directly targets the EGFR pathway;
* Prior severe infusion reaction to a monoclonal antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940 (Actual)
Dates: Start 2005-11; Primary Completion 2011-01 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rosenthal, MD, Principal Investigator — M.D. Anderson Cancer Center; Phuc Felix Nguyen-Tan, MD, Study Chair — CHUM Hospital Notre Dame
Locations (372):
- United States (363):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Providence Cancer Center, Anchorage, Alaska
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Auburn Radiation Oncology, Auburn, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Valley Medical Oncology, Fremont, California
  - Virginia K. Crosson Cancer Center at St. Jude Medical Center, Fullerton, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - San Francisco General Hospital Medical Center, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Stanford Cancer Center, Stanford, California
  - General Robert Huyser Cancer Center at David Grant Medical Center, Travis Air Force Base, California
  - Solano Radiation Oncology Center, Vacaville, California
  - Sutter Solano Medical Center, Vallejo, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Radiation Oncology, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Integrated Community Oncology Network at Southside Cancer Center, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Bay Medical, Panama City, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Georgia Cancer Center for Excellence at Grady Memorial Hospital, Atlanta, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Good Shepherd Hospital, Barrington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Good Samaritan Cancer Care Center at Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint John's Cancer Center at Saint John's Medical Center, Anderson, Indiana
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Radiation Oncology Associates Southwest, Fort Wayne, Indiana
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - NSMC Cancer Center - Peabody, Peabody, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Cancer Institute of Cape Girardeau, LLC, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Independence Regional Health Center, Independence, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Dartmouth - Hitchcock Concord, Concord, New Hampshire
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Ocean Medical Center at Meridian Health, Brick, New Jersey
  - Princeton Radiation Oncology Center, Jamesburg, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University Medical Center at Princeton, Princeton, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - Maimonides Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - St. Vincent's Comprehensive Cancer Center - Manhattan, New York, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Cancer Centers of North Carolina - Raleigh, Raleigh, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Wilmed Radiation Oncology Services, Wilson, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Precision Radiotherapy at University Pointe, West Chester, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Dubs Cancer Center at Rogue Valley Medical Center, Medford, Oregon
  - Providence Cancer Center at PMCC, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Oregon Health and Science University Cancer Institute, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Upper Delaware Valley Cancer Center, Milford, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Harrington Cancer Center, Amarillo, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Norris Cotton Cancer Center - North, Saint Johnsbury, Vermont
  - INOVA Alexandria Hospital, Alexandria, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - St. Francis Hospital, Federal Way, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
- Canada (9):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan

REFERENCES:
- [Result] Ang KK, Zhang Q, Rosenthal DI, Nguyen-Tan PF, Sherman EJ, Weber RS, Galvin JM, Bonner JA, Harris J, El-Naggar AK, Gillison ML, Jordan RC, Konski AA, Thorstad WL, Trotti A, Beitler JJ, Garden AS, Spanos WJ, Yom SS, Axelrod RS. Randomized phase III trial of concurrent accelerated radiation plus cisplatin with or without cetuximab for stage III to IV head and neck carcinoma: RTOG 0522. J Clin Oncol. 2014 Sep 20;32(27):2940-50. doi: 10.1200/JCO.2013.53.5633. PMID 25154822
- [Result] Truong MT, Zhang Q, Rosenthal DI, List M, Axelrod R, Sherman E, Weber R, Nguyen-Tan PF, El-Naggar A, Konski A, Galvin J, Schwartz D, Trotti A, Silverman C, Singh A, Godette K, Bonner JA, Jones CU, Garden AS, Shenouda G, Matthiesen C, Le QT, Bruner D. Quality of Life and Performance Status From a Substudy Conducted Within a Prospective Phase 3 Randomized Trial of Concurrent Accelerated Radiation Plus Cisplatin With or Without Cetuximab for Locally Advanced Head and Neck Carcinoma: NRG Oncology Radiation Therapy Oncology Group 0522. Int J Radiat Oncol Biol Phys. 2017 Mar 15;97(4):687-699. doi: 10.1016/j.ijrobp.2016.08.003. Epub 2016 Aug 12. PMID 27727066
- [Result] Schwartz DL, Harris J, Yao M, Rosenthal DI, Opanowski A, Levering A, Ang KK, Trotti AM, Garden AS, Jones CU, Harari P, Foote R, Holland J, Zhang Q, Le QT. Metabolic tumor volume as a prognostic imaging-based biomarker for head-and-neck cancer: pilot results from Radiation Therapy Oncology Group protocol 0522. Int J Radiat Oncol Biol Phys. 2015 Mar 15;91(4):721-9. doi: 10.1016/j.ijrobp.2014.12.023. PMID 25752384
- [Derived] Gharzai LA, Morris E, Schipper MJ, Kidwell KM, Nguyen-Tan PF, Rosenthal DI, Gillison ML, Jordan RC, Garden AS, Koyfman SA, Caudell JJ, Blakaj DM, Dunlap NE, Krempl GA, Longo JM, Jones CU, Gensheimer MF, Galloway TJ, DeMora L, Le QT, Shah JL, Suresh K, Mierzwa M. Treatment Interruption and Outcomes in Head and Neck Cancer: A Secondary Analysis of 3 Randomized Clinical Trials. JAMA Otolaryngol Head Neck Surg. 2025 Dec 4:e254203. doi: 10.1001/jamaoto.2025.4203. Online ahead of print. PMID 41343184
- [Derived] Caudell JJ, Torres-Saavedra PA, Rosenthal DI, Axelrod RS, Nguyen-Tan PF, Sherman EJ, Weber RS, Galvin JM, El-Naggar AK, Konski AA, Echevarria MI, Dunlap NE, Shenouda G, Singh AK, Beitler JJ, Garsa A, Bonner JA, Garden AS, Algan O, Harris J, Le QT. Long-Term Update of NRG/RTOG 0522: A Randomized Phase 3 Trial of Concurrent Radiation and Cisplatin With or Without Cetuximab in Locoregionally Advanced Head and Neck Cancer. Int J Radiat Oncol Biol Phys. 2023 Jul 1;116(3):533-543. doi: 10.1016/j.ijrobp.2022.12.015. Epub 2022 Dec 19. PMID 36549347
- [Derived] Mell LK, Shen H, Nguyen-Tan PF, Rosenthal DI, Zakeri K, Vitzthum LK, Frank SJ, Schiff PB, Trotti AM 3rd, Bonner JA, Jones CU, Yom SS, Thorstad WL, Wong SJ, Shenouda G, Ridge JA, Zhang QE, Le QT. Nomogram to Predict the Benefit of Intensive Treatment for Locoregionally Advanced Head and Neck Cancer. Clin Cancer Res. 2019 Dec 1;25(23):7078-7088. doi: 10.1158/1078-0432.CCR-19-1832. Epub 2019 Aug 16. PMID 31420360
- [Derived] Beitler JJ, Switchenko JM, Dignam JJ, McDonald MW, Saba NF, Shin DM, Magliocca KR, Cassidy RJ, El-Deiry MW, Patel MR, Steuer CE, Xiao C, Hudgins PA, Aiken AH, Curran WJ Jr, Le QT. Smoking, age, nodal disease, T stage, p16 status, and risk of distant metastases in patients with squamous cell cancer of the oropharynx. Cancer. 2019 Mar 1;125(5):704-711. doi: 10.1002/cncr.31820. Epub 2018 Dec 11. PMID 30548235
- [Derived] Weidhaas JB, Harris J, Schaue D, Chen AM, Chin R, Axelrod R, El-Naggar AK, Singh AK, Galloway TJ, Raben D, Wang D, Matthiesen C, Avizonis VN, Manon RR, Yumen O, Nguyen-Tan PF, Trotti A, Skinner H, Zhang Q, Ferris RL, Sidransky D, Chung CH. The KRAS-Variant and Cetuximab Response in Head and Neck Squamous Cell Cancer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2017 Apr 1;3(4):483-491. doi: 10.1001/jamaoncol.2016.5478. PMID 28006059
- Available data/document: Individual Participant Data Set: NCT00265941 — https://nctn-data-archive.nci.nih.gov/ — Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RT + Cisplatin | RT + Cisplatin + Cetuximab
Started | 470 | 470
Completed | 447 (Subjects with data available for the primary analysis are considered to have completed the study.) | 444 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 23 | 26
Not completed — Protocol Violation | 22 | 25
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients with follow-up
Groups:
- Total: Total of all reporting groups
Arm/Group | RT + Cisplatin | RT + Cisplatin + Cetuximab | Total
Number analyzed (Participants) | 447 | 444 | 891
Age, Continuous [Median (Full Range); unit: years] | 57 [31 to 79] | 58 [34 to 76] | 57 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 45 | 105
  Male | 387 | 399 | 786

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) (3-year Rate Reported)
Description: Progression-free survival (PFS) is defined as time from randomization to date of local, regional, or distant disease progression, or death from any cause. Patients last known to be alive without progression are censored at the date of last contact. Three-year rates were estimated by the Kaplan-Meier method. Local or regional progression is defined as an estimated increase in the size of the tumor (product of the perpendicular diameters of the two largest dimensions) of greater than 25%, taking as reference the smallest value of all previous measurements or appearance of new areas of malignant disease. Distant progression is defined as clear evidence of distant metastases.
Time Frame: From randomization until 434 failures have occurred, approximately 5 years from start of study. (Patients are followed until death or study termination, whichever occurs first.)
Population: Randomized eligible patients with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT + Cisplatin | RT + Cisplatin + Cetuximab
Number analyzed (Participants) | 447 | 444
percentage of participants | 61.2 [56.7 to 65.8] | 58.9 [54.2 to 63.6]
Statistical Analysis 1: Comparison: RT + Cisplatin vs RT + Cisplatin + Cetuximab; A total of 945 patients were required (900 analyzable) to test for a 25% reduction in the hazard associated with progression-free survival with 84% statistical power using a one-sided log-rank test at the 0.025 significance level (0.0238 after 3 interim analyses); Test type: Superiority; p = 0.76, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.88 to 1.32] — Reference arm = RT + cisplatin

2. Secondary Outcome: Overall Survival (OS) (3-year Rate Reported)
Description: Overall survival is defined as time from randomization to date of death from any cause. Patients last known to be alive are censored at the date of last contact. Three-year rates were estimated by the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Randomized eligible patients with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT + Cisplatin | RT + Cisplatin + Cetuximab
Number analyzed (Participants) | 447 | 444
percentage of participants | 72.9 [68.7 to 77.1] | 75.8 [71.7 to 79.9]
Statistical Analysis 1: Comparison: RT + Cisplatin vs RT + Cisplatin + Cetuximab; Arms were compared using a one-sided log-rank test at the 0.025 significance level; Test type: Superiority; p = 0.32, Log Rank; One-sided log-rank significance level of 0.025; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.74 to 1.21] — Reference level = RT + cisplatin

3. Secondary Outcome: Local-regional Failure (LRF) (3-year Rate Reported)
Description: Local-regional failure is defined as time from randomization to date of failure (local or regional progression), or distant disease progression, or death from any cause. Patients last known to be alive without progression are censored at the date of last contact. Distant disease progression is considered a competing risk. Local or regional progression is defined as an estimated increase in the size of the tumor (product of the perpendicular diameters of the two largest dimensions) of greater than 25%, taking as reference the smallest value of all previous measurements or appearance of new areas of malignant disease. Distant progression is defined as clear evidence of distant metastases. Three-year rates were estimated by the cumulative incidence method.
Time Frame: as for outcome 1
Population: Randomized eligible patients with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT + Cisplatin | RT + Cisplatin + Cetuximab
Number analyzed (Participants) | 447 | 444
percentage of participants | 19.9 [16.2 to 23.7] | 25.9 [21.7 to 30.1]
Statistical Analysis 1: Comparison: RT + Cisplatin vs RT + Cisplatin + Cetuximab; Test type: Superiority; p = 0.97, Log Rank; One-sided significance level of 0.025; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.99 to 1.70] — Reference level = RT + cisplatin

4. Secondary Outcome: Rate of Mucositis Toxicity ≥ Grade 3
Description: Grade 3 or higher Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 radiation mucositis definitely, probably, or possibly related to protocol treatment. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: From start of treatment until 434 failures have occurred, approximately 5 years from start of study. (Patients are followed until death or study termination, whichever occurs first.)
Population: Randomized eligible patients with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT + Cisplatin | RT + Cisplatin + Cetuximab
Number analyzed (Participants) | 447 | 444
percentage of participants | 33.3 [29.0 to 37.7] | 43.2 [38.6 to 47.9]

5. Secondary Outcome: Rate of Other Toxicity ≥ Grade 3 (Not Mucositis)
Description: Grade 3 or higher Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 other than radiation mucositis definitely, probably, or possibly related to protocol treatment. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: as for outcome 4
Population: Randomized eligible patients with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT + Cisplatin | RT + Cisplatin + Cetuximab
Number analyzed (Participants) | 447 | 444
percentage of participants | 89.3 [86.4 to 92.1] | 91.9 [89.4 to 94.4]

6. Secondary Outcome: Rate of Patients Who Tolerated Treatment
Description: A patient was considered to have tolerated treatment if radiation therapy was scored as per protocol or with acceptable variation, they received 2 cycles of cisplatin, and for arm 2, they received the initial dose of cetuximab and at least 5 weekly doses of cetuximab .
Time Frame: From start of treatment to end of treatment (6-7 weeks)
Population: Randomized eligible patients with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT + Cisplatin | RT + Cisplatin + Cetuximab
Number analyzed (Participants) | 447 | 444
percentage of participants | 84.8 [81.5 to 88.1] | 70.7 [66.5 to 75.0]

7. Secondary Outcome: Rate of Deaths ≤ 30 Days After Discontinuation of Protocol Treatment
Description: Patients who died during treatment or within 30 days after the end of treatment
Time Frame: From start of treatment to 30 days after the end of treatment
Population: Randomized eligible patients with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT + Cisplatin | RT + Cisplatin + Cetuximab
Number analyzed (Participants) | 447 | 444
percentage of participants | 1.8 [0.6 to 3.0] | 2.0 [0.7 to 3.3]

8. Secondary Outcome: Quality of Life as Measured by European Quality of Life Questionnaire (EQ-5D)
Description: The EQ-5D is a 2-part self-assessment questionnaire. First part is 5 items (mobility, self care, usual activities, pain/discomfort, anxiety/depression) each with 3 problem levels (1-none, 2-moderate, 3-extreme). Health states are defined by the combination of the leveled responses to the 5 dimensions, generating 243 health states to which unconsciousness and death are added. The 2nd part is a visual analogue scale (VAS) valuing current health state, measured on a 20-cm 10-point interval scale. Worst imaginable health state is scored as 0 at the bottom of the scale, and best imaginable health state is scored as 100 at the top. Both the 5-item index score and the VAS score are transformed into a utility score between 0 (worst health state) and 1 (best health state).
Time Frame: 3 months and 12 months
Population: Randomized eligible patients with EQ-5D data at the given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RT + Cisplatin | RT + Cisplatin + Cetuximab
Number analyzed (Participants) | 447 | 444
units on a scale
  EQ-5D 3 months: number analyzed (Participants) | 316 | 289
  EQ-5D 3 months | 0.78 (0.18) | 0.77 (0.15)
  EQ-5D 12 months: number analyzed (Participants) | 243 | 253
  EQ-5D 12 months | 0.84 (0.17) | 0.84 (0.16)
Statistical Analysis 1: Comparison: RT + Cisplatin vs RT + Cisplatin + Cetuximab; 3 months; Test type: Superiority; p = 0.74, Kolmogorov-Smirnov; 2-sided significance level of 0.05
Statistical Analysis 2: Comparison: RT + Cisplatin vs RT + Cisplatin + Cetuximab; 12 months; Test type: Superiority; p = 0.99, Kolmogorov-Smirnov; 2-sided significance level of 0.05

9. Secondary Outcome: Quality of Life as Measured by Proportion of Patients With Performance Status Scale for Head and Neck Cancer (PSS-HN) Scores ≤ 50
Description: The PSS-HN is a clinician rated instrument consisting of assessment of three functions (subscales): Normalcy of Diet, Eating in Public, and Understandability of Speech. The interviewer rates the patient on each scale based on the patient's responses to targeted questions. Scores on each subscale range from 0-100, with higher scores indicating better performance. It has been demonstrated to be reliable and valid in head and neck cancer patients.The site research nurse or clinical research associate (CRA) will determine the score on each of the subscales by performing a clinical evaluation and unstructured interview format. The PSS-HN takes approximately 5 minutes to complete.
Time Frame: 3 months and 12 months
Population: Randomized eligible patients with PSS-HN data at the given time point.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | RT + Cisplatin | RT + Cisplatin + Cetuximab
Number analyzed (Participants) | 447 | 444
proportion of participants
  Normalcy of Diet 3 months: number analyzed (Participants) | 282 | 272
  Normalcy of Diet 3 months | 0.80 [0.75 to 0.84] | 0.85 [0.80 to 0.89]
  Normalcy of Diet 12 months: number analyzed (Participants) | 234 | 223
  Normalcy of Diet 12 months | 0.37 [0.31 to 0.43] | 0.37 [0.31 to 0.44]
  Public Eating 3 months: number analyzed (Participants) | 283 | 272
  Public Eating 3 months | 0.62 [0.56 to 0.67] | 0.63 [0.59 to 0.67]
  Public Eating 12 months: number analyzed (Participants) | 234 | 230
  Public Eating 12 months | 0.18 [0.13 to 0.23] | 0.23 [0.18 to 0.28]
  Understandability of Speech 3 months: number analyzed (Participants) | 294 | 277
  Understandability of Speech 3 months | 0.09 [0.06 to 0.12] | 0.08 [0.05 to 0.12]
  Understandability of Speech 12 months: number analyzed (Participants) | 238 | 231
  Understandability of Speech 12 months | 0.05 [0.02 to 0.08] | 0.04 [0.02 to 0.07]
Statistical Analysis 1: Comparison: RT + Cisplatin vs RT + Cisplatin + Cetuximab; Diet 3-month; Test type: Superiority; p = 0.13, Chi-squared; 2-sided significance level of 0.05
Statistical Analysis 2: Comparison: RT + Cisplatin vs RT + Cisplatin + Cetuximab; Diet 12-month; Test type: Superiority; p = 0.87, Chi-squared; 2-sided significance level 0.05
Statistical Analysis 3: Comparison: RT + Cisplatin vs RT + Cisplatin + Cetuximab; Eating 3-month; Test type: Superiority; p = 0.39, Chi-squared; 2-sided significance level of 0.05
Statistical Analysis 4: Comparison: RT + Cisplatin vs RT + Cisplatin + Cetuximab; Eating 12-month; Test type: Superiority; p = 0.16, Chi-squared; 2-sided significance level of 0.05
Statistical Analysis 5: Comparison: RT + Cisplatin vs RT + Cisplatin + Cetuximab; Speech 3-month; Test type: Superiority; p = 0.81, Chi-squared; 2-sided significance level of 0.05
Statistical Analysis 6: Comparison: RT + Cisplatin vs RT + Cisplatin + Cetuximab; Speech 12-month; Test type: Superiority; p = 0.67, Chi-squared; 2-sided significance level of 0.05

10. Secondary Outcome: Quality of Life as Measured by Change From Baseline in Functional Assessment of Cancer Therapy-General (FACT-HN) at 12 Months
Description: The Functional Assessment of Cancer Therapy-Head and Neck (FACT-HN) is a 10-item self-report instrument designed to measure multidimensional quality of life in patients with head and neck cancer. It is to be administered with the FACT-General. There are 5 responses options, with 0=Not a lot and 4=Very much. All items are added together to obtain a total score which ranges from 0-40. Certain items must be reversed before it is added by subtracting the response from 4. It requires at least 50% of the items to be completed while the overall response rate of the FACT-HN including the FACT-G must be greater than 80%. If items are missing, the subscale scores can be prorated. A higher score indicated better QOL. Change from baseline to 12 months (12 months - baseline) is reported.
Time Frame: Baseline and 12 months
Population: Randomized eligible patients with baseline and 12-month FACT-HN data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RT + Cisplatin | RT + Cisplatin + Cetuximab
Number analyzed (Participants) | 229 | 226
units on a scale | -0.41 (18.9) | -5.11 (22.5)
Statistical Analysis 1: Comparison: RT + Cisplatin vs RT + Cisplatin + Cetuximab; Test type: Superiority; p = 0.016, t-test, 2 sided; 2-sided significance level of 0.05

11. Secondary Outcome: Correlation of Expression of Epidermal Growth Factor Receptor (EGFR) With PFS, OS, and LRF
Description: EGFR expression is categorized as high (>/=80%) and low (<80%) in order to compare outcome by favorable and unfavorable risk group, per protocol. Times are measured from randomization. Overall survival is defined as time from randomization to date of death from any cause. PFS is time to loco-regional progression (LRP), distant disease progression (DDP), or death. LRF is time to LRP, DDP, or death, with DDP considered a competing risk. Patients last known to be alive without event are censored at the date of last contact. LRP is defined as an estimated increase in the size of the tumor (product of the perpendicular diameters of the two largest dimensions) of greater than 25%, taking as reference the smallest value of all previous measurements or appearance of new areas of malignant disease. DDP is defined as clear evidence of distant metastases. Three-year LRF rates were estimated by the cumulative incidence method. Three-year PFS and OS rates were estimated by the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Randomized eligible patients with follow-up and EGFR data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Low EGFR: Less than 80% EGFR
- High EGFR: Greater than or equal to 80% EGFR
Arm/Group | Low EGFR | High EGFR
Number analyzed (Participants) | 235 | 145
percentage of participants
  Progression-free survival (PFS) | 63.5 [56.9 to 69.4] | 60.3 [51.7 to 67.8]
  Overall survival (OS) | 76.7 [70.6 to 81.7] | 75.0 [66.9 to 81.4]
  Loco-regional failure (LRF) | 21.7 [16.6 to 27.3] | 19.2 [13.1 to 26.1]
Statistical Analysis 1: Comparison: Low EGFR vs High EGFR; Progression-free survival is compared between favorable risk and unfavorable risk groups; Test type: Superiority; p = 0.60, Log Rank; 2-sided significance level = 0.05; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.79 to 1.51] — Reference level = low EGFR
Statistical Analysis 2: Comparison: Low EGFR vs High EGFR; Overall survival is compared between favorable risk and unfavorable risk groups; Test type: Superiority; p = 0.37, Log Rank; 2-sided significance level = 0.05; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.81 to 1.76] — Reference level = low EGFR
Statistical Analysis 3: Comparison: Low EGFR vs High EGFR; Local-regional failure; Test type: Superiority; p = 0.76, Log Rank; 2-sided significance level = 0.05; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.60 to 1.46] — Reference level = low EGFR

12. Secondary Outcome: Correlation of Pre-treatment Positron Emission Tomography (PET)/CT Maximum Standardized Uptake Value (SUVmax) With PFS, OS, and LRF
Description: SUVmax is categorized as high (>median) and low (</=median). All times are measured from randomization. Overall survival is defined as time from randomization to date of death from any cause. PFS is time to loco-regional failure (LRP), distant disease progression (DDP), or death. LRF is time to LRP, DDP, or death, with DDP considered a competing risk. Patients last known to be alive without event are censored at the date of last contact. LRP is defined as an estimated increase in the size of the tumor (product of the perpendicular diameters of the two largest dimensions) of greater than 25%, taking as reference the smallest value of all previous measurements or appearance of new areas of malignant disease. DDP is defined as clear evidence of distant metastases. Three-year LRF rates were estimated by the cumulative incidence method. Three-year PFS and OS rates were estimated by the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Randomized eligible N2-3 patients with follow-up and PET data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Low PET SUVmax: Less than or equal to median pretreatment PET SUVmax
- High PET SUVmax: Greater than median pretreatment PET SUVmax
Arm/Group | Low PET SUVmax | High PET SUVmax
Number analyzed (Participants) | 34 | 34
percentage of participants
  Progression-free Survival (PFS) | 55.9 [37.8 to 70.6] | 85.3 [68.2 to 93.6]
  Overall Survival (OS) | 85.3 [68.2 to 93.6] | 91.2 [75.1 to 97.1]
  Loco-regional failure (LRF) | 32.4 [17.4 to 48.3] | 11.8 [3.6 to 25.1]
Statistical Analysis 1: Comparison: Low PET SUVmax vs High PET SUVmax; Progression-free survival is compared between low and high SUVmax groups; Test type: Superiority; p = 0.01, Log Rank; 2-sided significance level = 0.05; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.12 to 0.75] — Reference level = low
Statistical Analysis 2: Comparison: Low PET SUVmax vs High PET SUVmax; Overall survival (OS) is compared between low and high SUVmax groups; Test type: Superiority; p = 0.10, Log Rank; 2-sided significance level = 0.05; Hazard Ratio (HR) = 0.38, 95% CI 2-sided [0.12 to 1.20] — Reference level = low
Statistical Analysis 3: Comparison: Low PET SUVmax vs High PET SUVmax; Loco-regional control (LRC) is compared between low and high SUVmax groups; Test type: Superiority; p = 0.04, Log Rank; 2-sided significance level = 0.05; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.10 to 0.97] — Reference level = low

13. Secondary Outcome: 2-year Nodal Relapse Rates in Clinical N2-3 Patients by Post-treatment PET/CT Finding and Nodal Response
Description: Patients are grouped by the combination of clinical nodal response status and the post-treatment PET/CT finding (negative or positive). Nodal relapse rate is calculated for each group by the cumulative incidence method. Relapse is defined as reappearance of tumor after complete response. If possible, relapse should be confirmed by biopsy.
Time Frame: From randomization to 2 years
Population: Randomized eligible N2-3 patients with follow-up and PET data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Clinical CR + Negative PET: Clinical nodal complete response; negative post-treatment PET/CT scan
- No Clinical CR + Negative PET: Did not have clinical nodal complete response; negative post-treatment PET/CT scan
- Clinical CR + Positive PET: Clinical nodal complete response; positive post-treatment PET/CT scan
- No Clinical CR + Positive PET: No clinical nodal complete response; positive post-treatment PET/CT scan
Arm/Group | Clinical CR + Negative PET | No Clinical CR + Negative PET | Clinical CR + Positive PET | No Clinical CR + Positive PET
Number analyzed (Participants) | 26 | 15 | 12 | 9
percentage of participants | 3.9 [0 to 11.4] | 33.3 [8.4 to 58.3] | 16.7 [0 to 38.8] | 11.1 [0 to 33.1]

ADVERSE EVENTS:
Description: Randomized eligible patients with follow-up data are included. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | RT + Cisplatin | RT + Cisplatin + Cetuximab
Serious Adverse Events (participants affected / at risk) | 208/447 | 237/444
Other Adverse Events (participants affected / at risk) | 442/447 | 433/444
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RT + Cisplatin (N=447) | RT + Cisplatin + Cetuximab (N=444)
Blood/bone marrow - Other (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 31 | 24
Hemoglobin (Blood and lymphatic system disorders) | 24 | 32
Hemolysis NOS (Blood and lymphatic system disorders) | 0 | 2
Arrhythmia NOS (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 1 | 1
Cardiac general - Other (Cardiac disorders) | 0 | 1
Cor pulmonale NOS (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 2
Myocardial ischemia (Cardiac disorders) | 3 | 5
Sinus arrhythmia (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 2 | 1
Otitis externa NOS (Ear and labyrinth disorders) | 1 | 0
Pain: External ear (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Endocrine - Other (Endocrine disorders) | 1 | 0
Abdominal distention (Gastrointestinal disorders) | 1 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 3 | 8
Constipation (Gastrointestinal disorders) | 10 | 14
Diarrhea NOS (Gastrointestinal disorders) | 7 | 14
Dry mouth (Gastrointestinal disorders) | 5 | 9
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 51 | 46
Enteritis necroticans (Gastrointestinal disorders) | 1 | 0
Esophageal pain (Gastrointestinal disorders) | 1 | 3
Esophageal perforation (Gastrointestinal disorders) | 1 | 0
Esophageal stenosis acquired (Gastrointestinal disorders) | 1 | 0
Esophagitis NOS (Gastrointestinal disorders) | 4 | 7
Fistula, GI: Abdomen NOS (Gastrointestinal disorders) | 0 | 1
Fistula, GI: Oral cavity (Gastrointestinal disorders) | 1 | 0
Fistula, Pulmonary/upper respiratory: Oral cavity (Gastrointestinal disorders) | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 2 | 0
Gastritis NOS (Gastrointestinal disorders) | 0 | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 2 | 3
Hemorrhage, GI: Upper GI NOS (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Intra-abdominal hemorrhage NOS (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Malabsorption (Gastrointestinal disorders) | 1 | 0
Mucositis/stomatitis (clinical exam): Anus (Gastrointestinal disorders) | 2 | 0
Mucositis/stomatitis (functional/symptomatic): Esophagus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 36 | 59
Oral pain (Gastrointestinal disorders) | 16 | 18
Pancreatitis NOS (Gastrointestinal disorders) | 1 | 0
Radiation mucositis (Gastrointestinal disorders) | 28 | 52
Rectal perforation (Gastrointestinal disorders) | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Salivary gland disorder NOS (Gastrointestinal disorders) | 2 | 5
Small intestinal stricture NOS (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 4 | 5
Tooth disorder NOS (Gastrointestinal disorders) | 1 | 0
Vomiting NOS (Gastrointestinal disorders) | 31 | 45
Chest pain (General disorders) | 1 | 2
Constitutional Symptoms - Other (General disorders) | 3 | 0
Death NOS (General disorders) | 1 | 3
Disease progression NOS (General disorders) | 0 | 1
Edema: head and neck (General disorders) | 2 | 0
Edema: limb (General disorders) | 0 | 2
Edema: trunk/genital (General disorders) | 0 | 1
Facial pain (General disorders) | 1 | 2
Fatigue (General disorders) | 8 | 27
Multi-organ failure (General disorders) | 0 | 3
Pain - Other (General disorders) | 4 | 2
Pain NOS (General disorders) | 1 | 0
Pyrexia (General disorders) | 12 | 28
Rigors (General disorders) | 4 | 4
Sudden death (General disorders) | 2 | 2
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1
Hypersensitivity NOS (Immune system disorders) | 0 | 15
Abdominal infection (Infections and infestations) | 0 | 2
Ano-rectal infection NOS (Infections and infestations) | 1 | 0
Bladder infection NOS (Infections and infestations) | 2 | 1
Bone infection NOS (Infections and infestations) | 2 | 1
Bronchitis NOS (Infections and infestations) | 0 | 1
Gingival infection (Infections and infestations) | 1 | 1
Implant site infection (Infections and infestations) | 2 | 0
Infection - Other (Infections and infestations) | 2 | 5
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Abdomen NOS (Infections and infestations) | 1 | 2
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Bladder (urinary) (Infections and infestations) | 1 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Blood (Infections and infestations) | 1 | 3
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Bone (osteomyelitis) (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Brain + Spinal cord (encephalomyelitis) (Infections and infestations) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Catheter-related (Infections and infestations) | 3 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Dental-tooth (Infections and infestations) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Esophagus (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Foreign body (e.g., graft, implant, pro (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Lung (pneumonia) (Infections and infestations) | 2 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Middle ear (otitis media) (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Mucosa (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Nose (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Oral cavity-gums (gingivitis) (Infections and infestations) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Pancreas (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Stomach (Infections and infestations) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Trachea (Infections and infestations) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Wound (Infections and infestations) | 3 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Blood (Infections and infestations) | 3 | 6
Infection with normal ANC or Grade 1 or 2 neutrophils: Catheter-related (Infections and infestations) | 0 | 3
Infection with normal ANC or Grade 1 or 2 neutrophils: Esophagus (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Larynx (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Lip/perioral (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Neck NOS (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Salivary gland (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Wound (Infections and infestations) | 1 | 1
Infection with unknown ANC: Lung (pneumonia) (Infections and infestations) | 1 | 3
Infection with unknown ANC: Trachea (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Opportunisitic infection (Infections and infestations) | 1 | 4
Otitis media NOS (Infections and infestations) | 1 | 0
Peritoneal infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia NOS (Infections and infestations) | 11 | 6
Respiratory tract infection NOS (Infections and infestations) | 1 | 1
Sepsis NOS (Infections and infestations) | 2 | 2
Skin infection (Infections and infestations) | 2 | 7
Urinary tract infection NOS (Infections and infestations) | 2 | 1
Wound infection (Infections and infestations) | 0 | 1
Burn (Injury, poisoning and procedural complications) | 1 | 0
Culture wound negative (Injury, poisoning and procedural complications) | 1 | 1
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 5 | 4
Hemorrhage, Pulmonary/upper respiratory: Trachea (Injury, poisoning and procedural complications) | 1 | 0
Radiation recall syndrome (Injury, poisoning and procedural complications) | 2 | 17
Tracheal stenosis (Injury, poisoning and procedural complications) | 0 | 2
Vascular access NOS complication (Injury, poisoning and procedural complications) | 3 | 2
Vessel injury-artery: Carotid (Injury, poisoning and procedural complications) | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 6
Aspartate aminotransferase increased (Investigations) | 3 | 6
Blood alkaline phosphatase increased (Investigations) | 1 | 3
Blood amylase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 5
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 20 | 19
Coagulopathy (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Inappropriate antidiuretic hormone secretion (Investigations) | 1 | 1
Leukopenia NOS (Investigations) | 34 | 38
Lipase increased (Investigations) | 1 | 0
Lymphopenia (Investigations) | 10 | 26
Metabolic/laboratory - Other (Investigations) | 0 | 3
Neutrophil count (Investigations) | 31 | 34
Platelet count decreased (Investigations) | 7 | 13
Prothrombin time prolonged (Investigations) | 1 | 0
Troponin I increased (Investigations) | 3 | 2
Troponin T increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 21 | 18
Anorexia (Metabolism and nutrition disorders) | 12 | 17
Blood iron increased (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 68 | 80
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia NOS (Metabolism and nutrition disorders) | 8 | 10
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 2 | 3
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 | 17
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 16
Hypoglycemia NOS (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 11 | 25
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 18
Hyponatremia (Metabolism and nutrition disorders) | 15 | 32
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 7 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Soft tissue necrosis: Head (Musculoskeletal and connective tissue disorders) | 1 | 2
Soft tissue necrosis: Neck (Musculoskeletal and connective tissue disorders) | 2 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1
Secondary Malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral ischemia (Nervous system disorders) | 2 | 2
Cognitive disorder (Nervous system disorders) | 0 | 1
Convulsions NOS (Nervous system disorders) | 0 | 2
Depressed level of consciousness (Nervous system disorders) | 6 | 1
Dizziness (Nervous system disorders) | 2 | 3
Dysgeusia (Nervous system disorders) | 1 | 4
Headache (Nervous system disorders) | 0 | 2
Hemorrhagic stroke (Nervous system disorders) | 0 | 2
Memory impairment (Nervous system disorders) | 1 | 1
Mental status changes (Nervous system disorders) | 0 | 2
Neuralgia NOS (Nervous system disorders) | 5 | 0
Neurology - Other (Nervous system disorders) | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1
Speech disorder (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 4
Syncope vasovagal (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 5 | 7
Depression (Psychiatric disorders) | 0 | 4
Insomnia (Psychiatric disorders) | 1 | 1
Psychosis aggravated (Psychiatric disorders) | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 1 | 0
Glomerular filtration rate (Renal and urinary disorders) | 1 | 0
Renal failure NOS (Renal and urinary disorders) | 17 | 12
Renal/genitourinary - Other (Renal and urinary disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hemorrhage, Pulmonary/upper respiratory: Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemorrhage, Pulmonary/upper respiratory: Pharynx (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Laryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Laryngeal stensos (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Laryngitis NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Mucositis/stomatitis (clinical exam): Larynx (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Mucositis/stomatitis (clinical exam): Pharynx (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Mucositis/stomatitis (functional/symptomatic): Larynx (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Mucositis/stomatitis (functional/symptomatic): Pharynx (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstruction/stenosis of airway: Pharynx (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary/upper respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne NOS (Skin and subcutaneous tissue disorders) | 0 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 2 | 10
Dermatology/skin - Other (Skin and subcutaneous tissue disorders) | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Nail disorder NOS (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fibrosis (Skin and subcutaneous tissue disorders) | 3 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0
Ulceration (Skin and subcutaneous tissue disorders) | 1 | 1
Hemorrhage/bleeding - Other (Vascular disorders) | 1 | 2
Hypertension NOS (Vascular disorders) | 0 | 1
Hypotension NOS (Vascular disorders) | 9 | 16
Peripheral ischemia (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 4 | 8
Vascular - Other (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RT + Cisplatin (N=447) | RT + Cisplatin + Cetuximab (N=444)
Blood/bone marrow - Other (Blood and lymphatic system disorders) | 31 | 31
Hemoglobin (Blood and lymphatic system disorders) | 262 | 250
Ear pain (Ear and labyrinth disorders) | 35 | 33
Hearing impaired (Ear and labyrinth disorders) | 127 | 114
Tinnitus (Ear and labyrinth disorders) | 117 | 106
Hypothyroidism (Endocrine disorders) | 82 | 70
Abdominal pain NOS (Gastrointestinal disorders) | 25 | 32
Constipation (Gastrointestinal disorders) | 170 | 146
Diarrhea NOS (Gastrointestinal disorders) | 76 | 92
Dry mouth (Gastrointestinal disorders) | 352 | 344
Dyspepsia (Gastrointestinal disorders) | 52 | 50
Dysphagia (Gastrointestinal disorders) | 431 | 415
Esophageal stenosis acquired (Gastrointestinal disorders) | 28 | 35
Esophagitis NOS (Gastrointestinal disorders) | 19 | 26
Gastrointestinal - Other (Gastrointestinal disorders) | 55 | 51
Nausea (Gastrointestinal disorders) | 252 | 243
Oral pain (Gastrointestinal disorders) | 143 | 158
Radiation mucositis (Gastrointestinal disorders) | 349 | 364
Salivary gland disorder NOS (Gastrointestinal disorders) | 179 | 159
Tooth disorder NOS (Gastrointestinal disorders) | 39 | 33
Vomiting NOS (Gastrointestinal disorders) | 170 | 179
Edema: head and neck (General disorders) | 119 | 117
Edema: limb (General disorders) | 23 | 19
Fatigue (General disorders) | 323 | 316
Pain - Other (General disorders) | 64 | 69
Pain NOS (General disorders) | 27 | 28
Pyrexia (General disorders) | 56 | 73
Rigors (General disorders) | 18 | 30
Gingival infection (Infections and infestations) | 25 | 23
Infection - Other (Infections and infestations) | 21 | 38
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 264 | 229
Radiation recall syndrome (Injury, poisoning and procedural complications) | 129 | 200
Alanine aminotransferase increased (Investigations) | 85 | 96
Aspartate aminotransferase increased (Investigations) | 71 | 69
Blood alkaline phosphatase increased (Investigations) | 48 | 34
Blood bilirubin increased (Investigations) | 17 | 38
Blood creatinine increased (Investigations) | 108 | 81
Leukopenia NOS (Investigations) | 207 | 206
Lymphopenia (Investigations) | 98 | 87
Metabolic/laboratory - Other (Investigations) | 46 | 46
Neutrophil count (Investigations) | 134 | 124
Platelet count decreased (Investigations) | 100 | 108
Weight decreased (Investigations) | 253 | 263
Anorexia (Metabolism and nutrition disorders) | 163 | 160
Dehydration (Metabolism and nutrition disorders) | 118 | 104
Hyperglycemia NOS (Metabolism and nutrition disorders) | 149 | 170
Hyperkalemia (Metabolism and nutrition disorders) | 40 | 46
Hypermagnesemia (Metabolism and nutrition disorders) | 29 | 17
Hypoalbuminemia (Metabolism and nutrition disorders) | 127 | 137
Hypocalcemia (Metabolism and nutrition disorders) | 90 | 116
Hypokalemia (Metabolism and nutrition disorders) | 84 | 102
Hypomagnesemia (Metabolism and nutrition disorders) | 106 | 152
Hyponatremia (Metabolism and nutrition disorders) | 165 | 186
Back pain (Musculoskeletal and connective tissue disorders) | 28 | 20
Fibrosis-deep connective tissue (Musculoskeletal and connective tissue disorders) | 23 | 21
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 23 | 31
Musculoskeletal/soft tissue - Other (Musculoskeletal and connective tissue disorders) | 33 | 48
Neck pain (Musculoskeletal and connective tissue disorders) | 80 | 96
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 46 | 44
Trismus (Musculoskeletal and connective tissue disorders) | 97 | 99
Dizziness (Nervous system disorders) | 43 | 55
Dysgeusia (Nervous system disorders) | 245 | 240
Headache (Nervous system disorders) | 56 | 83
Neuralgia NOS (Nervous system disorders) | 94 | 87
Peripheral motor neuropathy (Nervous system disorders) | 21 | 29
Peripheral sensory neuropathy (Nervous system disorders) | 110 | 121
Anxiety (Psychiatric disorders) | 64 | 48
Depression (Psychiatric disorders) | 64 | 62
Insomnia (Psychiatric disorders) | 68 | 72
Aspiration (Respiratory, thoracic and mediastinal disorders) | 31 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 110 | 94
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 60 | 65
Hiccups (Respiratory, thoracic and mediastinal disorders) | 24 | 20
Laryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 23 | 13
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 209 | 200
Laryngitis NOS (Respiratory, thoracic and mediastinal disorders) | 177 | 152
Mucositis/stomatitis (clinical exam): Larynx (Respiratory, thoracic and mediastinal disorders) | 85 | 74
Mucositis/stomatitis (clinical exam): Pharynx (Respiratory, thoracic and mediastinal disorders) | 240 | 218
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 185 | 154
Pulmonary/upper respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 47 | 36
Acne NOS (Skin and subcutaneous tissue disorders) | 13 | 291
Alopecia (Skin and subcutaneous tissue disorders) | 94 | 90
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 58 | 206
Dermatology/skin - Other (Skin and subcutaneous tissue disorders) | 150 | 158
Dry skin (Skin and subcutaneous tissue disorders) | 26 | 36
Pruritus (Skin and subcutaneous tissue disorders) | 34 | 153
Skin fibrosis (Skin and subcutaneous tissue disorders) | 220 | 213
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 94 | 87
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 26 | 28
Telangiectasia (Skin and subcutaneous tissue disorders) | 37 | 32
Hypotension NOS (Vascular disorders) | 31 | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.